CLINICAL TRIAL: NCT04589936
Title: Prone Position to Improve Oxygenation in COVID-19 Patients Outside Critical Care (PRONE-COVID Study)
Brief Title: Prone Position to Improve Oxygenation in COVID-19 Patients Outside Critical Care
Acronym: PRONE-COVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Jonathan Fuld, Consultant in Respiratory and Acute medicine, Cambridge University Hospitals NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 284061
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Pneumonia; Covid19
Keywords: Prone positioning; COVID-19; Pneumonia; Oxygenation
MeSH Terms: conditions — Pneumonia; COVID-19 | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: Case-control study design, with 1:1 for COVID-19 case versus pneumonia unrelated to COVID-19.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 (Experimental): Non-ventilated patients with COVID-19
  Interventions: Procedure: Prone positioning
- Pneumonia control (Active Comparator): Patients with pneumonia unrelated to COVID-19 requiring supplemental O2.
  Interventions: Procedure: Prone positioning

INTERVENTIONS:
Procedure: Prone positioning — Patient will first lay supine for a given time period, followed by lateral position on either side, then prone position, lastly return to supine position. Participants are anticipated to stay in prone position for a minimum of 30min to a maximum of 2 hours depending on tolerability. Participants will be guided in how to independently position themselves and rotate through the cycle of positions.
  Other Names: Proning

SUMMARY:
Prone positioning is known to improve the PaO2/FiO2 ratio and reduce mortality in patients with ARDS managed in the critical care setting. Therefore, it is incorporated into regular clinical practice of managing patients with ARDS in critical care and is being used as such in the COVID-19 outbreak. Given that prone positioning is recommended by the Intensive Care Society in non-ventilated patients with COVID-19, there is an urgent need to better understand the physiological effects of prone positioning in such cases. Furthermore, the translation and applicability of such a low-cost non-invasive intervention in a wider group of patients with pneumonia not specific to covid-19 infection, is an important consideration that merits investigation.

This single-centred observational study conducted at Cambridge University Hospitals NHS Foundation Trust aims to improve understanding of physiological effects of prone positioning in non-ventilated patients with COVID-19 and a control group of patients with non-COVID-19 related pneumonia. The study also aims to incorporate a small subset of patients, with an approximately even spread of COVID-19 and non-COVID cases, which allows for an additional exploratory descriptive report on prone positioning over a 24-hour period.

This study proposes that prone positioning improves oxygenation in non-ventilated patients with pneumonia (COVID-19 related or not) requiring supplemental oxygen managed outside of the critical care setting.

DETAILED DESCRIPTION:
COVID-19 (coronavirus disease 2019) caused by the infectious agent, SARS-CoV-2, was first recognised in Wuhan, Hubei Province, China in December 2019. Whilst a large proportion of COVID-19 illness within the community is mild, patients who are admitted to hospital with COVID-19 often have more severe disease and have a higher risk of developing COVID-19 complications including ARDS. Patients with ARDS are often managed on intensive care units that have evidence-based protocols for managing patients with ARDS. Prone positioning for such patients is a well-recognised component of ARDS critical care management. It is known to improve oxygenation and reduce oxygen requirements, as well as reduce mortality in patients with moderate to severe ARDS managed in critical care. The benefits of prone positioning as a technique to improve oxygenation in awake, non-intubated patients is less well-established. A few studies have showed prone positioning to be well-tolerated and improved oxygenation amongst non-intubated patients without respiratory support, as well as those requiring high-flow nasal oxygen or non-invasive ventilation support.

It remains unknown whether prone positioning is beneficial in patients with COVID-19 earlier in their disease, prior to requirement of non-invasive or invasive ventilation. This study therefore aims to better understand the physiological effects of prone positioning in patients with pneumonia with and without COVID-19.

This will be a single-centred interventional case-control study, comparing physiological effect of prone positioning in COVID-19 cases versus pneumonia unrelated to COVID-19. A sub-study of a smaller number of enrolled patients, with approximately even spread of COVID-19 and non-COVID cases, will allow an additional exploratory descriptive report on prone positioning over a 24-hour period.

Participant will be fitted with a Masimo monitoring device that enables continuous monitoring, and subsequent data storage and download of SpO2, heart rate, end tidal CO2 and respiratory rate. The sub-study investigating the effects of a longer duration of proning will involve applying a non-invasive positional sensor to automatically detect the participant's position, and correlate it with the patient's physiological parameters as well as tolerability. Qualitative data on patient's tolerability of prone positioning will also be collected.

It is anticipated that each participant will be their own control, enabling comparison of SpO2 in supine, lateral, prone and again supine positions. Summary statistics of mean, median, range, interquartile range, and range for each position for participants will be summarised. The data from the two arms will initially be analysed separately, then pooled to determine if a larger sample size impacts results. A multilevel regression model with average SpO2 as outcome will be fitted to assess the effect of lying position on SpO2. Additional models such as mixed models incorporating multiple repeated measurements/endpoints may be considered/fitted for exploratory analyses. Data from questionnaires will be reported by summary statistics where possible. Free text responses may be grouped into themes, and parametric or non-parametric tests will be used to analyse the VAS data further.

All data will be transferred into a Case Report Form (CRF) which will be anonymised. The investigator will obtain written informed consent from each participant before any study-specific activity is performed. Before the start of the study, or implementation of any amendment, we will obtain approval of the protocol, protocol amendments, informed consent forms and other relevant documents from the REC.

ELIGIBILITY:
Inclusion Criteria:

1. Have confirmed or suspected COVID-19 or non-COVID pneumonia (confirmed with radiological changes)
2. FiO2 ≥24% or requiring basic respiratory support (supplementary oxygen via face mask, nasal cannula, venturi, non-rebreathe bag) to achieve clinical target SpO2 (e.g. SpO2 92-96%), ensuring patient is on appropriately titrated oxygen to be within this range.
3. Be able to provide informed consent
4. Communicate and cooperate with the procedure
5. Rotate and adjust position independently
6. No anticipated airway issues

Exclusion Criteria:

The presence of any of the following will mean participants are ineligible:

1. Signs of respiratory distress (e.g. respiratory rate ≥35, accessory muscle use)
2. Immediate need for intubation
3. Haemodynamic instability or new arrhythmia
4. Unstable spine/thoracic injury/recent abdominal surgery
5. Pregnancy (2nd/3rd trimester)
6. At risk of pressure sores/ulcers
7. Neurological issues-frequent seizures
8. Facial injury that would make prone position difficult
9. Gastrointestinal issues-frequent vomiting or diarrhoea that would make prone position difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Peripheral Oxygen saturation | 1 year (June 2021)
  Oxygenation measured by peripheral saturations in relation to inspired oxygen (FiO2) when patient is prone versus a supine or lateral position using a Masimo device

SECONDARY OUTCOMES:
PaO2 :FiO2 ratio calculated from formulae | 1 year (June 2021)
  To evaluate effects of prone position versus supine or lateral position on derived measures of oxygenation (Pa02:Fi02 ratio calculated from formulae) in relation to inspired oxygen.
Respiratory rate measured with Masimo device | 1 year (June 2021)
  Effects of prone versus supine or lateral position on respiratory rate
Heart rate measured with Masimo device | 1 year (June 2021)
  Effects of prone versus supine or lateral position on heart rate
Blood pressure measured with Masimo device | 1 year (June 2021)
  Effects of prone versus supine or lateral position on blood pressure
Patient reported severity of breathlessness on a continuous linear scale of 0 to 10cm (10cm being the most severe) | 1 year (June 2021)
  To evaluate whether prone position reduces patient reported severity of breathlessness assessed by visual assessment score.
Patient tolerability of prone position on a continuous linear scale of 0 to 10cm (10cm being the most unacceptable) | 1 year (June 2021)
  To evaluate patient tolerability of prone position assessed by visual assessment score.
Investigator experience of delivering prone positioning | 1 year (June 2021)
  To evaluate investigator experience of delivering prone positioning in this study by free text question responses.
To assess patient's peripheral oxygen saturation | 1 year (June 2021)
  To evaluate the natural position of patients (with the aid of position sensors) who are encouraged to position themselves prone over a 24-hour period (which include sleep) and relationship with oxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Fuld, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elharrar X, Trigui Y, Dols AM, Touchon F, Martinez S, Prud'homme E, Papazian L. Use of Prone Positioning in Nonintubated Patients With COVID-19 and Hypoxemic Acute Respiratory Failure. JAMA. 2020 Jun 9;323(22):2336-2338. doi: 10.1001/jama.2020.8255. PMID 32412581